CLINICAL TRIAL: NCT03915041
Title: Effects of tDCS Combined With Virtual Reality on Anxious Ruminations in Healthy Subjects With a Vulnerability to Rumination
Brief Title: Effects of tDCS Combined With VR on Anxious Ruminations in Healthy Subjects With a Vulnerability to Rumination
Acronym: REVISTIM-XX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: RC17_0390
Record Dates: First submitted 2019-02-18; First posted 2019-04-16 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Rumination
Keywords: virtual reality; brain stimulation; tDCS; phenomenology
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR + active brain stimulation (Experimental): Exposure to a virtual reality world with active transcranial electric stimulation
  Interventions: Device: VR + active brain stimulation
- VR + sham brain stimulation (Sham Comparator): Exposure to a virtual reality world with sham transcranial electric stimulation
  Interventions: Device: VR +sham brain stimulation

INTERVENTIONS:
Device: VR + active brain stimulation — Active Brain stimulation (tDCS) is applied during exposition to virtual reality (20 minutes)
  Arms: VR + active brain stimulation
Device: VR +sham brain stimulation — Sham Brain stimulation (tDCS) is applied during exposition to virtual reality (20 minutes)
  Arms: VR + sham brain stimulation

SUMMARY:
This study proposes: to evaluate 1) whether the combination of virtual reality (VR) and active tDCS provides better rumination attenuation than the combination of VR and tDCS placebo 2) the acceptability and experiential experience of combining these two well known medical devices.

DETAILED DESCRIPTION:
Inclusion visit:

* Confirmation of eligibility criteria
* Written informed consent

Visit 1 and 2 (or end of study visit) :

Before first ruminations induction :

* Completion of Brief State Rumination Inventory (BSRI), State-Trait Anxiety (STAI), Inventory, Visual Analogic Scale (VAS), Ruminative Response Scale - Short Form (RRS-SF), Beck depression Inventory (BDI)
* EEG recording

Then Procedure for inducing ruminations using a pre-recorded voice listened to in an audio headset alternating statements promoting a positive, neutral and negative introspection and self-judgment attitude (the latter are heard at the end to initiate the rumination process) over 8 minutes

Then

* Completion of Brief State Rumination Inventory (BSRI), Inventory, Visual Analogic Scale (VAS), Beck depression Inventory (BDI),
* EEG recording
* Pulse and blood pressure measurements

Then immersion in a relaxing virtual environment for 20 minutes with active or sham placebo.

• Cutaneous conductance measurement and eye-tracking during immersion

At the end of immersion :

* Completion of Brief State Rumination Inventory (BSRI), Inventory, Visual Analogic Scale (VAS), Beck depression Inventory (BDI), IGroup presence questionnaire (IPQ)
* Pulse and blood pressure measurements

Then again procedure for inducing ruminations .

At the end of ruminations induction :

* Completion of Brief State Rumination Inventory (BSRI), State-Trait Anxiety (STAI), Inventory, Visual Analogic Scale (VAS), Beck depression Inventory (BDI), tolerance questionnaires
* Debriefing

ELIGIBILITY:
Inclusion Criteria:

* Without any particular ethnic and psychosocial criteria
* Subject to ruminations (personality trait) documented by a RRS-SF score >30
* Subjects with score to BDI scal <14 assessed during first visit
* Subjects without psychiatric or addictive disorders.
* Subjects who do not meet all the diagnostic criteria for an anxiety disorder or characterized depressive episode.

Exclusion Criteria:

* contraindication to tDCS (neurosurgical history, intracranial device, skin problems)
* current virtual reality intolerance
* history of psychiatric or addictive disorders
* Use of psychotropic drugs
* Use of non psychotropic treatments significantly influencing mood or level of anxiety
* pregnant or breast-feeding women
* Neurological pathology, locomotor disability, or sensory (vestibular, visual, auditory ...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Change in anxious ruminations after anodal tDCS and virtual reality | within 1 week
  Change in anxious ruminations after anodal tDCS and virtual reality will be evaluated to compare the effects of tDCS associated with virtual reality versus virtual reality alone (+ tDCS placebo) to reduce ruminations.
  Evaluate with Brief State Ruminative Inventory (BSRI). It is a scale with 8 items. Each item is VAS with a score ranging between 0 and 100. The total score is sum of each item score (Total /800)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No